CLINICAL TRIAL: NCT00488969
Title: Effectiveness of Controlled-Release Morphine for Chronic Neuropathic Pain After Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas N. Bryce, MD, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H133N060027; GCO # 90-135
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Neuropathic Pain; Spinal Cord Injury
Keywords: Morphine; Chronic Pain; Spinal Cord Injury; Neuropathic Pain
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified-release morphine then Placebo (Active Comparator): up to a ceiling dose of 120 mg
  Interventions: Drug: Modified-release morphine; Drug: Placebo
- Placebo then modified-release morphine (Placebo Comparator): Matching placebo
  Interventions: Drug: Modified-release morphine; Drug: Placebo

INTERVENTIONS:
Drug: Modified-release morphine — During the first three weeks of each treatment (drug or placebo), the dose will be escalated toward a maximally tolerated dose or a dose sufficient to eliminate pain (up to a ceiling dose of 120 mg), whichever is reached first. During the entire fourth and fifth week of each period, subjects will receive their maximally tolerated dose of study medication. During the sixth and seventh weeks, they will undergo a seven-day dose tapering and a seven-day complete washout of the study drug.
  Other Names: Modified-release morphine sulfate
Drug: Placebo

SUMMARY:
We would like to learn if a medicine called "modified-release morphine sulfate" (Avinza) helps reduce Spinal Cord Injury (SCI)-related pain that has lasted a long time. "Modified-release" means that the medicine in the capsules is slowly released to the body, instead of being released all at once. Avinza is approved by the Food and Drug Administration for the treatment of pain, but we do not know how effective Avinza is in reducing SCI-related pain.

DETAILED DESCRIPTION:
Neuropathic pain occurs as a result of damage to neural tissue either in the peripheral or in the central nervous system. Three types of neuropathic pain after SCI are especially difficult to treat: at level central pain (ALCP), at level radicular pain (ALRP), and below level central pain (BLCP). Various analgesic medications with distinct mechanisms and sites of action are currently used in clinical practice for treatment of neuropathic pain after SCI, including antidepressants, anticonvulsants, nonsteroidal anti-inflammatory drugs (NSAIDs), and opioids. These analgesic medications, when evaluated in animal models of SCI pain and in the treatment of other neuropathic pain states, have been shown to have only modest pain reducing effect. This modest effect is seen clinically as the majority of persons with SCI receiving these drugs continue to experience pain, which is severe and disabling in one third of cases.

This study proposes to examine the efficacy of oral modified release morphine in reducing pain in persons with neuropathic pain after SCI who have not adequately responded to other oral pharmacologic, psychologic, or physical interventions. Only subjects who have failed prior pain treatment regimes will be enrolled. Failure of pain regimen is defined as the presence of pain in spite of medication(s) or other pain treatment, such as biofeedback or other psychological or physical therapy interventions prescribed by a physician.

The following hypothesis will be tested: morphine, when added to non-opioid medications, is more effective than placebo in reducing pain and increasing activity and subjective well-being, in persons with ALCP, ALRP and BLCP. In order to test this hypothesis, a randomized, double blind, placebo-controlled, two period cross-over trial is proposed, during which subjects with ALCP, ALRP, and BLCP will receive daily placebo or modified release morphine while being closely monitored and assessed for: (1) adverse effects, (2) quality and intensity of pain, (3) intensity of allodynia and hyperalgesia, and (4) activity levels and well-being.

All subjects whether assigned to the placebo or active drug will be able to continue any previously prescribed or non-prescribed (over-the-counter) non-opioid medication that has been taken on a regular basis, without dose change, for at least three weeks prior to study entry. These medications may include but are not limited to the analgesics: acetaminophen and any non-steroidal anti-inflammatory drugs; local anesthetics- topical patches such as the lidocaine patch or otherwise; and adjuvant pain medications of the anti-depressant or anticonvulsant classes. Subjects will not be allowed to take any opioid medication, including non-opioid-opioid combination analgesics, other than the study drug for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65
* Diagnosis of traumatic spinal cord injury
* Neuropathic pain (pain related to the nervous system) rated at least 4 on a 11-point numeric rating scale at the time of screening
* Pain classified as at level radicular pain (ALRP), at level central pain (ALCP) or below level central pain (BLCP).
* Pain that is present regularly for at least 3 months prior to enrollment, in spite of medication or other pain treatment. This pain can be paroxysmal in nature (attacks of pain).
* Ability to understand instructions and reliably provide pain assessments
* Willingness to stop current opioid medications, if any
* If a female with childbearing potential, using an approved method of birth control (intrauterine device (IUD), barrier protection, a contraceptive implantation system or injection (Norplant® or Depo-Provera®), oral contraceptive pills, or celibacy)

Exclusion Criteria:

* A known sensitivity to opioids
* A history of substance or alcohol abuse within the past 2 years
* A need for elective surgery involving preoperative or postoperative analgesics or anesthetics during the study period
* Other chronic pain that cannot be differentiated from ALCP, ALRP, or BLCP
* A history of active cancer, excluding basal carcinoma of the skin, in the past 3 years
* Serum creatinine levels >= 2.5 mg/dl or hepatic (liver) dysfunction with serum ALT, AST, GGT, or total bilirubin >= 3 times the upper limit of normal
* Participation in any drug study in the last three months
* Currently pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pain severity | Average of daily ratings over 14 days
  Pain severity rated using a 0-10 Numeric Rating Scale (NRS)

SECONDARY OUTCOMES:
Short McGill Pain Questionnaire (modified) (SF-McGill) | up to 14 weeks
Opioids cognitive effects scale | up to 14 weeks
Patient Generated Index for activity (PGI) | up to 14 weeks
Daily number of attacks of paroxysmal pain | up to 14 weeks
Quantitative sensory testing | up to 14 weeks
  Allodynia, hyperalgesia, and temporal summation (determined using quantitative sensory testing)
Subject global impression of change | up to 14 weeks
Short-Form 36 (SF-36) | up to 14 weeks
Positive And Negative Affect Schedule (PANAS) | up to 14 weeks
Brief Patient Health Questionnaire (PHQ-9) | up to 14 weeks
Multidimensional Pain Inventory Life Interference subscale (MPI-LIS) | up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bryce, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States